CLINICAL TRIAL: NCT06262724
Title: Reliability of Chest Wall Perforator Flaps for Breast Reshaping Following Massive Weight Loss
Brief Title: Breast Reshaping Following Massive Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perforator Flaps
Record Dates: First submitted 2024-01-22; First posted 2024-02-16 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Ptosis

STUDY DESIGN:
Intervention Model Description: All patients were subjected to the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery (Other): Surgical intervention for breast reshaping utilizing chest wall perforators for auto-augmentation.
  Interventions: Procedure: Breast auto-augmentation

INTERVENTIONS:
Procedure: Breast auto-augmentation — Single group assignment. All patients included were subjected to utilizing chest wall perforator flaps for breast reshaping.

SUMMARY:
Reliability of Chest Wall Perforator Flaps for Breast Reshaping following Massive Weight Loss

DETAILED DESCRIPTION:
Conditions for inclusion in the study:

* Ptotic and deflated breasts following massive weight loss (MWL) with Pittsburgh Rating Scale (PRS) score of 2-3 as described by Songet al. (Song AY, Jean RD, Hurwitz D, Fernstrom MH, Scott JA, Rubin JP. A Classification of Contour Deformities after Bariatric Weight Loss: The Pittsburgh Rating Scale. Plast Reconstr Surg. 2005;116:1535-1544).
* MWL is defined as loss of 50% or greater of excess weight, following surgical or non-surgical interventions.
* Stable weight for at least 6 months, to achieve metabolic and nutritional homeostasis and decrease the risk of surgical complications.
* Body mass index (BMI): 18.5 - 30 kg/m2.
* Patients seeking autologous augmentation or refusing implants.
* Patients requiring simultaneous contouring of lateral chest wall redundancy.

Exclusion Criteria:

* Weight fluctuations in the previous 6 months.
* Medical co-morbidities (e.g., uncontrolled diabetes, uncontrolled hypertension, thyroid diseases, hormonal disturbances, cardiopulmonary diseases).
* Hereditary conditions that affect wound healing (e.g., Ehler Danlos Syndrome, Progeria).
* Active smokers (Smokers are required to stop smoking 1 month before surgery).
* Nutritional deficiencies (e.g., iron, vitamin B12, protein, folate).
* Previous breast surgery.
* Congenital breast deformity (e.g., tuberous breasts).
* Breast masses.
* Pregnant or lactating patients.

Local breast examination:

* Skin dimpling and intertrigo.
* Masses.
* Axillary lymph nodes.
* Position of nipple areola complex (NAC) and degree of ptosis (Regnault classification).
* Parenchyma (PRS score)
* Skin laxity.
* Direct breast anthropometry (baseline measurements for comparison and to guide surgical intervention):

The following measurements were assessed as described by Quieregatto et al. (Quieregatto PR, Hochman B, Ferrara SF, Furtado F, Liebano R, Neto MS, Ferreira LM. Anthropometry of the Breast Region: How to Measure? Aesth Plast Surg. 2014; 38:344-349) to help in pre-operative planning and to be compared to post-operative results.

A. Anatomical landmarks:

1. AAL: Anterior axillary line
2. MCP: Mid-clavicular plane
3. MHP: Mid-humeral plane
4. N: Nipple
5. SN: Sternal notch
6. IMF: Inframammary fold

B. Linear measurements (using tape measure): (Ideal values described by Liu YJ, Thomson JG. Ideal Anthropomorphic Values of the Female Breast. Annals of Plastic Surgery. 2011;67(1), 7-11.):

1. SN-N (21 cm)
2. N-IMF (8 cm)
3. N-N (21 cm)

Photographic assessment:

Seven standardized digital photographs were taken with the following parameters: Fixed camera settings, identical background and lighting and a tape on the floor to ensure that patients stand in the same place and the same room (Swanson E. A Measurement System and Ideal Breast Shape. Evidence-Based Cosmetic Breast Surgery. Springer, Cham. 2017;19-31.):

1. Frontal view
2. Left lateral view.
3. Right lateral view.
4. A view with 45° rotation to the left.
5. A view with 45° rotation to the right.
6. Left lateral view with arms up.
7. Right lateral view with arms up.

Pre-operative mammography:

* To exclude pre-operative tumors, cysts, and fat necrosis.
* To assess pre-operative breast volume.
* To be compared to post-operative mammography.

Surgical technique:

1. Pinch test of excess tissue in the lateral chest wall (donor flap).
2. Mapping of the perforators by hand-held Doppler probe.
3. Mastopexy and auto-augmentation (as described by Rubin JP, Khachi G. Mastopexy After Massive Weight Loss: Dermal Suspension and Selective Auto-Augmentation. Clinics in Plastic Surgery. 2008;35(1), 123-129.), which includes Wise Pattern with preservation of inferior and central pedicle, in addition to lateral extension to encompass the lateral chest wall skin roll.
4. Intraoperative perforator marking (thoracodorsal artery perforator versus intercostal artery perforator).
5. Flap transposition and anchoring to the chest wall by permanent sutures to the periosteum of the second rib for auto-augmentation and filling of the upper pole.
6. Skin closure and surgical drains in the breast and donor site.
7. Wound dressing and surgical bra.
8. Post-operative follow-up: The patient was evaluated:

   * During the first 48 hours: for hematoma, NAC compromise and drain removal according to amount and color (less than 50 cc/ serous) and then discharged.
   * At postoperative day 7, 10, 14 and 21: to detect any complications such as seroma, wound dehiscence, infection (redness, hotness, tenderness, discharge).

Patient evaluation: Final results were documented at 6 and 12 months through:

1. Direct breast anthropometry: To compare to pre-operative measurements, as well as assess the sustainability of the post-operative results.
2. Mammography:

   * To measure breast volume.
   * For signs of fat necrosis (as described by Chala LF, de Barros N, de Camargo Moraes P, Endo E, Kim SJ, Pincerato KM, Carvalho FM, Cerri GG. Fat Necrosis of the Breast: Mammographic, Sonographic, Computed Tomography, and Magnetic Resonance Imaging Findings. Curr Probl Diagn Radiol. 2004;33(3):106-26.), which reflect partial or total flap loss:

   Oil cyst (radiolucent mass surrounded by a thin fibrous membrane). Fibrotic reaction (irregular spiculated density). Calcifications (thin-walled calcifications in oil cysts or coarse irregular calcifications with radiolucent areas interspersed between them).
3. Photographic assessment (as before):

The pre and post-operative photos were analyzed by three plastic surgery consultants who were not involved in the study, through a PowerPoint presentation. Data provided by surgeons were grouped under three categories: poor, good or excellent. The inter-observer concordance rate was statistically calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years old.
* Weight:

  * Loss of 50% or greater of excess weight, following surgical or non-surgical interventions (MWL).
  * Stable weight for at least 6 months, to achieve metabolic and nutritional homeostasis and decrease the risk of surgical complications (Rubin et al., 2004).
* BMI: 18.5 - 30 kg/m2.
* Ptotic and deflated breasts with Pittsburgh Rating Scale (PRS) score 2-3 (Song, et al., 2005).
* Patients seeking autologous augmentation or refusing implants.
* Patients requiring simultaneous contouring of lateral chest wall redundancy.

Exclusion Criteria:

* Weight fluctuations in the previous 6 months.
* Medical co-morbidities (e.g., uncontrolled diabetes, uncontrolled hypertension, thyroid diseases, hormonal disturbances, cardiopulmonary diseases).
* Hereditary conditions that affect wound healing (e.g., Ehler Danlos Syndrome, Progeria).
* Active smokers (Smokers are required to stop smoking 1 month before surgery).
* Nutritional deficiencies (e.g., iron, vitamin B12, protein, folate).
* Previous breast surgery.
* Congenital breast deformity (e.g., tuberous breasts).
* Breast masses.
* Pregnant or lactating patients.
* PRS score 1.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Measurement of breast volume by sono-mammography | One year follow-up
  Use of sono-mammography to measure the breast volume in cubic centimetres preoperatively, after 6 months and after one year following surgery. The equation used to measure the breast volume was as follows:
  Breast volume = π/4 × (W × H × C) where W = breast width, H = breast height, and C=compression thickness in craniocaudal mammography)

SECONDARY OUTCOMES:
Sternal notch to nipple distance | One-year follow-up
  Measures of the distance between sternal notch and nipple in centimetres in both sides using tape preoperatively, after 6 months and one year following surgery
Nipple to inframammary fold distance | One-year follow-up
  Measures of the distance between nipple and intramammary fold in centimetres in both sides using tape preoperatively, after 6 months and one year following surgery
Measure of nipple-to-nipple distance | One-year follow-up
  Measure of the distance between both nipples in centimetres using tape preoperatively, after 6 months and one year following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Amr AW Mabrouk, MD, Study Director — Faculty of Medicine, Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No